CLINICAL TRIAL: NCT01351662
Title: An Intervention to Reduce Psychosocial and Biological Indicators of Stress in African American Lupus Patients: The Balancing Lupus Experiences With Stress Strategies (BLESS) Study
Brief Title: Balancing Lupus Experiences With Stress Strategies
Acronym: BLESS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: BLESS
Record Dates: First submitted 2011-05-09; First posted 2011-05-11 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus; stress
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Self management program (Experimental): The Arthritis Self-Management Program (ASMP) will be administered to 15 African American lupus patients participating in an ongoing "SLE Clinic Database Project" at the Medical University of South Carolina (MUSC). Fifteen other patients will serve as controls and receive usual care.
  Interventions: Behavioral: Arthritis Self Management Program

INTERVENTIONS:
Behavioral: Arthritis Self Management Program — Intervention activities will consist of six weekly sessions of the Arthritis Self-Management Program (ASMP). Sessions will be administered in a group setting with the 15 African American lupus patients randomly assigned to the intervention arm of the study. Fifteen other patients will serve as controls and receive usual care. Patients participating in the stress intervention will receive six weeks of peer led sessions ranging in disease-specific and more general self-help content. The intervention will include homework assignments to practice and record use of session techniques and to complete worksheets regarding session-specific topics and activities. Usual care will include a brief explanation of the disease and relevant literature.

SUMMARY:
Linking a psychosocial stress intervention with clinical measures of stress in African American lupus patients will assess the utility of this method in reducing perceived stress, and provide the necessary preliminary steps toward future investigations of potential mechanisms.

DETAILED DESCRIPTION:
To begin to fill this research void, a stress intervention will be piloted and both biological specimens and questionnaire responses collected to assess changes in stress state following the intervention in patients who participated in the intervention compared to those who did not participate in the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* African American
* Diagnosis of Lupus

Exclusion Criteria:

* Previous participation in a disease self management program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Perceived stress | Four months
  Psychosocial stress will be assessed by five validated measures. The State-Trait Anxiety Inventory (STAI), The Perceptions of Racism Scale, modified version of the Medical Outcomes Study (MOS) health distress scale, adapted by the Stanford Patient Education Research Center, and The Beck Depression Inventory.
Biological Indicators of stress | Four months
  Salivary specimens will be collected immediately preceding intervention activities, immediately following intervention activities, and four months post-intervention activities for analyses of salivary cortisol and Dehydroepiandrosterone (DHEA). Specified markers were chosen because they are easy to collect, relatively inexpensive, and reliable measures of stress.

SECONDARY OUTCOMES:
Quality of Life | Four months
  Quality of life will be assessed using two instruments that describe a spectrum of quality of life outcomes; The LUP-QOL and the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F). Stanford Patient Education Research Center Questionnaires assessing medical outcomes will also be used. These scales also assess whether key behaviors concerning communicating with health care providers and health care utilization have changed.

CONTACTS AND LOCATIONS:
Overall Officials: Edith M Williams, PhD, Study Director — University of South Carolina; James C Oates, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States